CLINICAL TRIAL: NCT05455385
Title: The Added Value of a Third Supervised Training Session (Ground Exercises or Hydrotherapy) to a Standard 12-week Rehabilitation Program After Breast Cancer: Pilot Study
Brief Title: The Added Value of a Third Supervised Training Session to a Standard 12-week Rehabilitation Program After Breast Cancer: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: s63338
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: rehabilitation; hydrotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: 3-arm randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator)
  Interventions: Other: standard 12-week rehabilitation program
- Hydrotherapy group (Experimental)
  Interventions: Other: standard 12-week rehabilitation program; Other: extra session hydrotherapy
- Ground exercise group (Experimental)
  Interventions: Other: standard 12-week rehabilitation program; Other: extra session ground exercises

INTERVENTIONS:
Other: standard 12-week rehabilitation program — The standard program consisted of 1 session in the fitness room and 1 session in the sports hall/week during 12 weeks.
Other: extra session hydrotherapy — The hydrotherapy group receives 1.5h additional hydrotherapy/week in addition to the standard program.
  Arms: Hydrotherapy group
Other: extra session ground exercises — The ground exercise group, receives 1.5h ground exercises/week in addition to the standard program.
  Arms: Ground exercise group

SUMMARY:
Breast cancer is the most common type of cancer diagnosed in women. A good rehabilitation program is essential for a good recovery after breast cancer, both physically and mentally. The aim of this study is to determine if there is an added value of a third supervised training session within a standard 12-week rehabilitation program to improve physical and mental functioning after breast cancer. The investigators also want to determine the added value of hydrotherapy as a third training session within a 12-week rehabilitation program compared to a third training session with ground exercises to improve physical and mental functioning after breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* men and women after surgery for breast cancer (mastectomy/breast-conserving and/or axillary gland resection/sentinel biopsy)
* possible (neo)adjuvant chemotherapy and radiotherapy have been completed
* hormone and/or immunotherapy may still be ongoing

Exclusion Criteria:

* comorbidities that make hydrotherapy impossible, i.e. open wounds or allergy to chlorine
* oncological unstable disease
* terminal patients
* severe physical disabilities
* severe mental disabilities
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Shoulder mobility | 12 weeks
  Shoulder Range of Motion (ROM) is measured with a Dr. Rippstein Plurimeter-V analogue inclinometer
Arm volume | 12 weeks
  Arm circumference measurements are performed bilaterally using a perimeter, a flexible stainless-steel rod with a measuring tape attached every 4 cm and a 20 g weight at the end.Arm circumference is measured at the level of the olecranon and at 4, 8, 12, 16 and 20 cm proximal and distal to the olecranon. The volume of the arm is calculated using a formula. The relatively excessive arm volume is then calculated as follows: (volume of operated limb - volume of non-operated limb) / volume of non-operated limb) x 100.
Force based on handgrip strength | 12 weeks
  Handgrip strength is measured with the Jamar Handheld Dynamometer
Flexibility by means of the sit-and-reach test | 12 weeks
  The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back.
Exercise capacity based on 6-minute walk test | 12 weeks
  The 6-minute walk test is used to assess patients' gait pattern, walking speed and cardiorespiratory endurance. It measures the maximum distance the patient can comfortably cover in 6 minutes.
Body image using the Body Image Scale | 12 weeks
  The BIS is a patient-reported outcome measure to evaluate the body image during and after cancer treatment. The BIS consists of 10 items and measures cognitive, affective and behavioral symptoms of body image. It uses a 4-point scale, where 0 = not at all and 3 = very much. The total score ranges from 0 to 30 and can be calculated by adding the 10 items together. The higher the score, the higher the level of body image disturbance.
self-reported pain using the Brief Pain Inventory | 12 weeks
  The BPI measures the severity of pain symptoms and interference with daily functioning using an 11-point scale. It has 4 questions for pain (worst pain, least pain, average pain and pain right now) and 7 for pain-related functioning (general physical activity, mood, ability to walk, work and household tasks, relationships with others, sleep, vitality). The total score is calculated by averaging all the different questions. A higher score indicates a higher barrier
Fatigue using the Functional Assessment of Chronic Illness Therapy - Fatigue Scale | 12 weeks
  FACIT-F scale measures the impact of fatigue caused by the treatment of chronic diseases. It consists of 13 items, with a score between 13 and 65. A higher score on the scale indicates more fatigue
Anxiety and depression using the Hospital Anxiety and Depression Scale | 12 weeks
  The HADS measures core symptoms of anxiety and depression without including physical symptoms. It is a short questionnaire that is easy to use. It consists of an anxiety scale and a depression scale, both containing 7 items with a total score from 0-21 where the higher the score, the more complaints. A score higher than 8 can be an indication for a psychiatric condition
Quality of life using the McGill Quality Of Life questionnaire | 12 weeks
  The McGill Quality of Life Questionnaire measures multiple dimensions and overall quality of life of people with a life-threatening illness. It measures quality of life according to 5 domains: physical symptoms, physical well-being, psychological, existential and support. A scale of 0-10 is used for each question with anchors at each end. The scores consist of three parts: (1) Part "A" is a Single-Item Scale (MQOL-SIS) that measures overall quality of life, (2) five subscales discussed above, and (3) a total score that is the average of the five subscales. Before calculating the MQOL scores, the scores for items 1, 2, 3, 5, 6, 7, and 8 must be converted by subtracting the raw score for each item from 10. For the results we only look at the third part, namely the total score. A higher score means a better quality of life
Physical functioning using the Patient-Reported Outcomes Measurement Information System | 12 weeks
  The PROMIS-PF includes many questionnaires in the areas of physical, mental and social health that can be used in the general population and in individuals suffering from chronic conditions. In our study we use the PROMIS for Physical Functioning, which is a 5-point scale where 1 = effortless and 10 = impossible. The score range goes from 10 to 50. A higher PROMIS score represents more of the concept being measured. So the higher the score, the better the physical functioning
Patient Specific Complaints | 12 weeks
  The PSC can be used to gain insight into the activities that a patient has difficulty with because of his/her symptoms. The patient is asked to name three activities in which he/she experiences discomfort in daily life or has difficulty with because of his/her symptoms or condition, and that he/she would like to improve with the therapy. The selected activities are scored on the amount of effort it takes him/her to perform this activity on an 11-point scale, where 0 = no effort at all and 10 = impossible. The total score is calculated by averaging the three individual scores. The higher the score, the more problems are experienced in performing the actions
Global Perceived Effect | 12 weeks
  The GPE can be used to measure the patient's opinion of recovery. The GPE consists of 2 items that must be answered on a 7-point scale. The scale runs from fully recovered to worse than ever. The first item is about "To what extent have you recovered from your complaints since the start of the treatment?" where 7 = worse than ever and 0 = completely improved. The second item is about "How satisfied are you with your treatment?". This scale goes from 7 = absolutely dissatisfied and 0 = absolutely satisfied
Attendance: number of times the participant was present | 12 weeks
  By attendance we mean the number of times the participant was present during the rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: An De Groef, Prof, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium